CLINICAL TRIAL: NCT01776671
Title: Efficacy of Once Daily Gastroretentive Gabapentin (Gralise) in the Treatment of Post Amputation Pain
Brief Title: Once Daily Gabapentin in the Treatment of Post Amputation Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chicago Anesthesia Pain Specialists (Other)
Responsible Party: Principal Investigator, Kenneth D Candido, Chairman of the Anesthesia Department, Chicago Anesthesia Pain Specialists
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Advocate-IRB-5367
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Pain; Quality of Life
MeSH Terms: conditions — Pain | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gralise (Other): Efficacy of Gralise
  Interventions: Drug: Gralise

INTERVENTIONS:
Drug: Gralise — Titration starting 300 mg/day up to 1800 mg/day over 2 weeks

SUMMARY:
Phantom limb pain (PLP) is a common disorder reported by the patients who undergo amputation. Even though the cause of PLP remains unclear, Gabapentin has been widely used. The purpose of this study is to evaluate the accuracy and efficacy achieved in using of extended release Gabapentin. Reducing the incidence of chronic post-amputation pain and improving clinical outcomes postoperatively.

DETAILED DESCRIPTION:
Phantom limb pain (PLP) is a common disorder reported by the patients who undergo amputation from peripheral vascular disease, peripheral neuropathic disease, neoplasm or traumatic events. Even though the cause of PLP remains unclear and the large number of treatments has been suggested, there is no single treatment regimen proving long lasting pain relief for PLP. However Gabapentin is widely used and have been well suggested recently for the treatment of neuropathic pain.

The purpose of this study is to evaluate the accuracy and efficacy achieved in using of extended release Gabapentin to offer effective pain relief, improvement of sleep function, and decrease problematic side effects related to the peaks and valleys of the drug's short cycle in patients with PLP. Gabapentin has been clearly demonstrated to be effective in neuropathic pain and epilepsy, but as a treatment option for post amputation pain, it has not been tested.

Approximately, 20 patients will be enrolled in the study, after a titration of two weeks a changing in pain intensity and quality of life will be obtained at subsequent visits. We are expected that the accuracy will be of benefit in reducing the incidence of chronic post-amputation pain and improving clinical outcomes postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have post amputation pain persisting for more than six months.
* Be considered in reasonably good health, in the opinion of the investigator, other than the post amputation pain at the screening visit (based upon the results of the medical and surgical history, vital signs, pulse oximetry and physical examination.
* Be ≥ 18 years of age at the time of screening.
* Female subject are eligible only if all of the following apply:

  * Not pregnant ( negative serum pregnancy test at the screening visit);
  * Not lactating
  * Consented to use barrier contraceptive methods to avoid pregnancy beginning at least 10 days before check -in and continuing throughout the study up to month after the end of the study.
* Voluntarily provide written informed consent.
* Must in the investigator's opinion, to be able to comply with the study procedure.

Exclusion Criteria:

* Hypersensitivity or allergy to gabapentin
* History of co-existing epilepsy or uncontrolled seizure disorder
* Subject is suffering from dementia or any cognitive dysfunction
* Have an uncontrolled or poorly controlled major psychiatric condition (e.g. schizophrenia, major depression) or who have clinically significant anxiety or depression
* Severe cardiopulmonary or liver disease
* Impaired kidney function testing
* Patient receiving hemodialysis
* Subjects with current uncontrolled depression or other uncontrolled psychiatric disorder
* Subjects currently taking anticonvulsants for any reason of treatment
* History of untreated alcohol abuse
* History of gastrointestinal symptoms such as: diarrhea, dyspepsia or gastro duodenal ulcers
* Subjects with history of gastric reduction surgery
* Any other clinically significant condition, or unstable inter-current illness that would, in the opinion of the investigator, preclude study participation or interfere with the assessment of the pain
* Clinically significant of uncontrolled hypo or hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Numeric Rating Scale at rest | Visit 1, 2, 3, 4, 5, 6
  Visit 1, baseline; visit 2, one week after visit one; visit 3, two weeks after visit 1; visit 4, two weeks after visit 3; visit 5, six weeks after visit 3; visit 6, two weeks after visit 5.

SECONDARY OUTCOMES:
Change in Pain numeric rating scale at movement. | Visit 1, 2, 3, 4, 5, 6
  Visit 1, baseline; visit 2, one week after visit one; visit 3, two weeks after visit 1; visit 4, two weeks after visit 3; visit 5, six weeks after visit 3; visit 6, two weeks after visit 5.

OTHER OUTCOMES:
Modified brief pain inventory (short form) | Visit 1, and visit 5
  Visit 1, baseline; visit 5, eight weeks after visit 1.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Candido, M.D., Principal Investigator — Chicago Anesthesia Pain Specialists
Locations (1):
- Chicago Anesthesia Pain Specialists, Chicago, Illinois, United States